CLINICAL TRIAL: NCT04638946
Title: Optimizing Exercise for the Treatment of Anxiety
Brief Title: Exercise for Anxiety
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01348
Record Dates: First submitted 2020-11-02; First posted 2020-11-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titration to high intensity exercise (Experimental)
  Interventions: Behavioral: Titration to high intensity exercise (T-HIE)
- Low intensity exercise (Active Comparator)
  Interventions: Behavioral: Low intensity exercise prescription

INTERVENTIONS:
Behavioral: Titration to high intensity exercise (T-HIE) — All participants will receive psychoeducation regarding the rationale for using exercise as a strategy to create immediate changes in mood and anxiety. Participants will be instructed in basic motivational principles (e.g., breaking up goals into smaller parts, using rewards) based on information in Exercise for Mood and Anxiety. Participants will begin at low intensity with the goal of titrating to high intensity by 2 weeks prior to the end of trial (Week 6). If a participant achieves at least 70% of the duration goal at the target heart rate, he/she will be titrated to the next dose level (moderate intensity). This will continue until high intensity exercise is achieved. Prescription is based on heart rate reserve((maximum heart rate [220-age] - resting heart rate)*intensity percent - resting heart rate. Intensity percent lower/upper limits for moderate intensity are 40-59% and for high intensity are 60-84%.
  Arms: Titration to high intensity exercise
Behavioral: Low intensity exercise prescription — All participants will receive psychoeducation regarding the rationale for using exercise as a strategy to create immediate changes in mood and anxiety. Participants will be instructed in basic motivational principles (e.g., breaking up goals into smaller parts, using rewards) based on information in Exercise for Mood and Anxiety. Prescription is based on heart rate reserve ((maximum heart rate [220-age] - resting heart rate)*30-39% (lower/upper limit of zone) - resting heart rate.
  Arms: Low intensity exercise

SUMMARY:
90 sedentary adults with a primary anxiety disorder and high anxiety sensitivity will be randomized to either 8 weeks of 1) low intensity exercise, or 2) flexible titration to high intensity exercise (HIE). Blinded, validated clinician-rated and patient-rated outcomes will be assessed over treatment and at 1- and 3-month follow-up. To better understand what mechanisms influence decisions to exercise in the real-world, we will use of heart rate (HR) as an objective mechanistic target for exercise intensity, examine changes in valuation of exercise through a neuroeconomics task, examine changes in interoceptive sensitivity with a heartbeat detection task, and integrate of ecological momentary assessment (EMA) to measure effects of immediate changes in mood with exercise on anxiety outcomes and adherence.

ELIGIBILITY:
Inclusion Criteria

* Males and females ages 18-65
* Primary psychiatric diagnosis of generalized anxiety disorder (GAD), social anxiety disorder, or panic disorder
* Anxiety Sensitivity Index-3 score of ≥23 (i.e., high anxiety sensitivity)
* Currently sedentary (≤60 minutes of moderate intensity exercise per week for the past 3 months)
* Body mass index <40
* Able and willing to provide informed consent

Exclusion Criteria

* Lifetime history of Bipolar I or II or any psychotic disorder
* Bulimia or anorexia in the past 6 months
* Substance use disorder in the past 3 months
* Current PTSD (past PTSD is allowed)
* High current suicide risk (active suicidal ideation with plan and intent) as indicated by a score of ≥4 on the Columbia Suicide Severity Rating Scale (C-SSRS) consistent with a need for referral to higher level of care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety Sensitivity Index-3 (ASI-3) score | Baseline, Week 8
  The ASI-3 is an 18-item measure of fear of anxiety sensations with three subscales (physical, cognitive, social concerns). The total score ranges from 0 (lowest anxiety sensitivity) to 72 (highest anxiety sensitivity).
Change in Clinical Global Impressions/Severity Scale score | Baseline, Week 8
  A validated Clinical Global Impressions/Severity Scale (CGI) anchored for anxiety disorders measures overall functioning and clinical improvement. CGI-S is rated from 1 (least disordered) to 7 (most disordered).Scores of 1 or 2 on the CGI-I at post-treatment will represent significant response.

SECONDARY OUTCOMES:
Engagement | Week 12, Week 20
  Completion of exercise of any intensity (proportion of 75min assigned)
Adherence | Week 8, Week 12, Week 20
  Percentage of duration goals achieving target heart rate
Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A) Score | Week 1, Week 4, Week 8, Week 12, Week 20
  14-item clinician-rated measure of severity of anxiety symptoms; The total score ranges from 0 (least severe anxiety symptoms) to 56 (most severe anxiety symptoms).
Work and Social Adjustment Scale (WSAS) Score | Week 1, Week 4, Week 8, Week 12, Week 20
  5 item self-report scale measing impairment in functioning with total score ranging from 0 (no impairment) to 40 (severe impairment).
Overall Anxiety Severity and Impairment Scale (OASIS) Score | Week 1, Week 4, Week 8, Week 12, Week 20
  A 5-item self-report scale measuring anxiety symptom severity and impairment due to anxiety; response items are coded from 0 to 4 and can be summed to obtain a total score range from 0 (least severity and impairment) to 20 (most severity and impairment).
Multidimensional Assessment of Interoceptive Awareness (MAIA-2) Score | Week 1, Week 4, Week 8, Week 12, Week 20
  A 37-item measure with 8 subscales assessing noticing bodily sensations, not distracting from bodily sensations, not worry about bodily sensations, attention regulation, emotional awareness (awareness of connection between emotions and bodily sensations), self-regulation of distress by body sensations, body listening, and trusting one's body.
Score on Montgomery-Asberg Depression Rating Scale (MADRS) | Week 1, Week 4, Week 8, Week 12, Week 20
  A 10-item clinician-rated measure of depression severity. Total score ranges from 0 (normal/no symptoms) to 60 (severe depression).
7 Day Physical Activity Recall Questionnaire (PAR) Score | Weekly from Week 0 (screening) to Week 20
  interviewer-administered measure of self-reported weekly physical activity
Barriers Specific-Self-Efficacy Scale (BARSE) Score | Week 1, Week 4, Week 8, Week 12, Week 20
  13-item measure, will assess barriers to exercise and will be used as a covariate predicting exercise engagement
Physical Activity Enjoyment Scale (PACES) | Week 1, Week 4, Week 8, Week 12, Week 20
  18-item measure assessing enjoyment of exercise
Preferences for and Tolerance of the Intensity of Exercise Questionnaire (PRETIE-Q) Score | Week 1, Week 4, Week 8, Week 12, Week 20
  16-item measure assessing preferences for different exercise intensities, with strong ability to differentiate preferences for HIE vs. LIE.
Heartrate | Weekly from week 1 to week 20
  Measured by the Fitbit Charge 3
Ecological Momentary Assessment (EMA) Score | Weekly from week 1 to week 20
  Surveys will consist of five 0-100 Likert scale items assessing mood, anxiety, motivation, energy, and enjoyment.
Neuroeconomics willingness-to-pay (WTP) auction task adapted for exercise | Week 1, Week 4, Week 8, Week 12, Week 20
  will evaluate the subjective threshold between an option's anticipated value and its cost (maximum amount WTP for an expected outcome) and is based on the Becker-DeGroot-Marschak (BDM) auction task68, modified for exercise. Participants will have the opportunity to avoid exercising for a specific timeframe (e.g., 1min, 15min) at a specific intensity (low, moderate, high). The task will first be administered on paper (21-item questionnaire), which will be computerized in line with training aims.
Heartrate by Heartbeat Detection Task | Week 1, Week 4, Week 8, Week 12, Week 20
  Participants silently count their heartbeats for 6 trials of approximately 20-30 seconds (~5 minutes) while being monitored on an EKG to assess accuracy of reporting. This will assess interoceptive accuracy and will be used as a covariate at baseline and change with intervention will be assessed over time.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Szuhany, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to the PI

DOCUMENTS (1):
  • Informed Consent Form (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT04638946/ICF_000.pdf